CLINICAL TRIAL: NCT01704352
Title: Cognitive Behavioral Therapy for Insomnia in Euthymic Bipolar Disorder: a Randomized Controlled Trial
Brief Title: Cognitive Behavioral Therapy for Insomnia in Euthymic Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/1033
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Bipolar Disorder; Insomnia
Keywords: Cognitive Behavioral Therapy; CBT-I
MeSH Terms: conditions — Bipolar Disorder; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT-I (Active Comparator): Cognitive behavioral therapy for insomnia (CBT-I) is a multicomponent treatment consisting of sleep restriction therapy, psychoeducation about sleep, stimulus control, stabilizing circadian rhythm and challenging beliefs and perception of sleep.
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia
- Treatment as usual (No Intervention): Treatment as usual (TAU) consists of pharmacological and supportive psychosocial treatment according to the needs of the patient.

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for insomnia — CBT-I will be given during 3-6 sessions according to need by two therapists being either psychiatrists or psychologists with clinical experience in CBT-I.
  Arms: CBT-I

SUMMARY:
Patients with bipolar disorder suffer from sleep disturbances, even in euthymic phases. Changes in sleep are frequent signs of a new episode of (hypo)mania or depression. Cognitive behavioral therapy for insomnia is an effective treatment for primary insomnia, but has not been introduced to patients with bipolar disorder. The aim is to compare cognitive behavioral therapy added to 'treatment as usual' with just 'treatment as usual'. The investigators hypothesize that cognitive behavioral therapy will improve quality of sleep, stabilize minor mood variations and prevent new mood episodes in euthymic patients with bipolar disorder and insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling criteria for SCID-1-verified bipolar I or II disorder
* Euthymic, as defined by Montgomery Åsberg Depression Rating Scale (MADRS) not higher than eleven, and Young Mania Rating scale (YMRS) not higher than five.
* Fulfilling DSM-IV criteria for primary insomnia or insomnia related to another mental disorder, as assessed by the Insomnia Interview Schedule (IIS).

Exclusion Criteria:

* Being or having been in a defined affective episode the last month before inclusion
* Hospitalization in the last two months before inclusion
* Working night shifts
* Sleep apnea
* Medical conditions incompatible with participation.
* Inability to cooperate in the 3-week initial phase before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in quality of sleep at 8 weeks | At 8 weeks from randomization
  As assessed by the Insomnia Severity Index (ISI)
Change from baseline in quality of sleep at 6 months follow-up | 6 months from end of treatment phase
  As assessed by the Insomnia Severity Index (ISI)

SECONDARY OUTCOMES:
Variation in sleep registration from baseline to 8 weeks | At 8 weeks
  Comparing registrations of sleep by sleep diaries, actigraphs and polysomnography.
Variation in sleep registration from baseline to 6 months follow-up | At 6 months
  Comparing registrations of sleep by sleep diaries, actigraphs and polysomnography.

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Morken, PhD Prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Østmarka Psychiatric Department, St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Derived] Steinan MK, Krane-Gartiser K, Langsrud K, Sand T, Kallestad H, Morken G. Cognitive behavioral therapy for insomnia in euthymic bipolar disorder: study protocol for a randomized controlled trial. Trials. 2014 Jan 16;15:24. doi: 10.1186/1745-6215-15-24. PMID 24433249
- See also: Related Info — http://www.ntnu.no/sleep-bp